CLINICAL TRIAL: NCT01096940
Title: A Randomized, Open-label, 3-way Crossover Phase I Study in Type 2 Diabetes Mellitus Patients Treated With Metformin to Evaluate the Pharmacokinetics and Pharmacodynamics of Simvastatin During Coadministration With AZD1656 and to Evaluate the Pharmacokinetics of AZD1656 During Coadministration With Simvastatin
Brief Title: Study To Assess the Pharmacokinetics of AZD1656 During Coadministration With Simvastatin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: D1020C00029
Record Dates: First submitted 2010-03-30; First posted 2010-03-31 (Estimated); Last update posted 2010-11-08 (Estimated); Status verified 2010-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Glucose lowering
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — AZD1656; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): AZD1656
  Interventions: Drug: AZD1656
- 2 (Experimental): Simvastatin
  Interventions: Drug: simvastatin
- 3 (Experimental): AZD1656 + simvastatin
  Interventions: Drug: AZD1656; Drug: simvastatin

INTERVENTIONS:
Drug: AZD1656 — Oral tablet, BID dose
  Arms: 1; 3
Drug: simvastatin — Oral tablet, single dose
  Arms: 2; 3

SUMMARY:
To assess the pharmacokinetics of AZD1656 during coadministration with Simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of T2DM for at least 1 year, treated with any metformin or metformin with one other oral anti-diabetic drug (OAD)
* Body mass index between greater than or equal to 19 and less than or equal to 42 kg/m2
* HbA1c greater than 6.5% at enrollment

Exclusion Criteria:

* Clinically significant illness or clinically relevant trauma, as judged by the Investigator, within 2 weeks before the first administration of the IP
* Significant cardiovascular event within the last 6 months prior to enrollment (eg, myocardial infarction/acute coronary syndrome, revascularisation procedure, stroke or transient ischaemic attack) or heart failure New York Heart Association (NYHA) class III-IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of AZD1656 on the steady state pharmacokinetics of simvastatin (including simvastatin acid) and vice versa by assessment of AUC(0-24) and Cmax. | Frequent blood samples for PK analysis will be drawn during 24 hours post morning dose on day 4 in each treatment period (1-3)

SECONDARY OUTCOMES:
To evaluate the effect of AZD1656 on the steady state pharmacokinetics of simvastatin and simvastatin acid and vice versa by assessment of tmax, t1/2 and CL/F (only for AZD1656) | Frequent serial blood samples will be drawn during 24 hours post morning dose on Day 4 in each treatment period (1-3)
To evaluate the steady state pharmacokinetics of the AZD1656 metabolite when AZD1656 is administered with and without simvastatin, by assessment of AUC(0-24), Cmax and tmax. | Frequent serial blood samples will be drawn during 24 hours post morning dose on Day 4 in each treatment period (1-3)
To evaluate the effect of AZD1656 on the pharmacodynamics of simvastatin by assessment of AUC(0-t) and Cmax of active 3-hydroxy-3-methyl-glutaryl-CoA reductase inhibitors. | Frequent serial blood samples will be drawn during 24 hours post morning dose on Day 4 in each treatment period (1-3)
To evaluate the safety and tolerability of AZD1656 alone and in combination with simvastatin by assessments of adverse events, laboratory variables, electrocardiogram, blood pressure, pulse, results of physical examination, and weight. | At pre entry, during the study days,

CONTACTS AND LOCATIONS:
Overall Officials: Jolene K. Berg, MD, Principal Investigator — Cetero Research, Inc.; Stanko Skrtic, Study Director — AstraZeneca; Mirjana Kujacic, Study Chair — AstraZeneca
Locations (1):
- Research Site, San Antonio, Texas, United States